CLINICAL TRIAL: NCT04840303
Title: The Effectiveness and Cost-effectiveness of Mental Wellness Youth Hubs
Brief Title: The Effectiveness and Cost-effectiveness of Mental Wellness Youth Hub
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); The Boys' and Girls' Clubs Association of Hong Kong (Other); Caritas Medical Centre, Hong Kong (Other); Hong Kong Federation of Youth's Group (HKFYG) (Other); Hong Kong Playground Association (Unknown); Hong Kong Children and Youth Services (Unknown); St. James' Settlement (Other)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Chair Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 19-680
Record Dates: First submitted 2021-03-03; First posted 2021-04-12 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Mental Stress
Keywords: youth mental health
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hub user group (Experimental): This group receives community-based mental wellness youth hub services for young people to enhance personal strengths and overall mental well-being.
  Interventions: Behavioral: LevelMind@JC Mental Wellness Youth Hubs
- non-hub user active control group (No Intervention): This group does not receive the community-based mental wellness youth hub services but other generic youth services in the community.
- non-hub user community control group (No Intervention): This group does not receive any youth services in the community.

INTERVENTIONS:
Behavioral: LevelMind@JC Mental Wellness Youth Hubs — Mental Wellness Youth Hubs Intervention aims to set up a series of community-based hubs for young people to enhance cognitive abilities, personal strengths and overall mental well-being. Among the experimental group participants (hub users), they are further divided into three tiers according to their psychological distress level. Tier 1 are youths with mild psychological distress level, who will be invited to participate in some innovative and interesting youth projects and activities (e.g., board game and floral artistry). Tier 2 are youths who have moderate level of psychological distress, or at risk for mental illness. Trained social workers will offer them with specific interventions (e.g., CBT, sleep intervention) according to their needs. Tier 3 are youths with severe level of psychological distress who are at risk for mental disorders. Diagnostic and medical assessment services will be delivered by psychiatrist or clinical psychologists.
  Arms: Hub user group

SUMMARY:
The proposed study is to be carried out with 6000-7000 youths aged 12 - 24 in Hong Kong. The purpose of the study is to investigate the effectiveness and cost-effectiveness of a Hub project for young people: LevelMind@JC. This study is conducted by LevelMind@JC in collaboration with partnering NGOs including the Boys' & Girls' Clubs Association of Hong Kong (BGCA), Caritas Hong Kong, Hong Kong Federation of Youth's Group (HKFYG), Hong Kong Playground Association (HKPA), Hong Kong Children and Youth Services (HKCYS) and St James' Settlement (SJS). It is a 1-year quasi experimental controlled study which aims to examine if these hubs can enhance young people's cognitive abilities, personal strengths and overall mental well-being. 1800 participants would be recruited, including 600 Hub users, 600 non-hub users (but receiving services from participating NGOs), and 600 community youth not receiving any youth services. Participants will be assessed at baseline and follow-ups (e.g., 3 months, 6 months, and 12 months); completing questionnaires and answering questions during a 3- hour interview. Hub users with mild to moderate mental distress will receive different psychological treatments according to their needs. For youths who are at risk for mental disorders, diagnostic and medical assessment services will be delivered by psychiatrists or clinical psychologists. Findings will allow us to better understand the effectiveness of this kind of community-based hubs for young people, improve mental wellness training of youth social workers; and in a long run, develop a community-based support model that is sustainable, scalable and replicable.

ELIGIBILITY:
Inclusion Criteria:

* For hub-user group (experimental group): 12 - 24 year- old hub users who receive community-based mental wellness youth hub services for young people.
* For non-hub user group (active control group): 12 -24 year- old youths who do not receive the community-based mental wellness youth hub services but other generic youth services in the community.
* For non-hub user group (passive control group): 12 -24 year- old community youth who do not receive any youth services in the community.

Exclusion Criteria:

* Youths with known diagnosis of psychiatric disorders (including Depression, Generalized Anxiety Disorder, Panic Disorder, Phobia, Obsessive Compulsive Disorder, Bipolar Disorder, Eating Disorder, Personality Disorder, Post-Traumatic Stress Disorder and Psychotic Disorder)
* Youths who receive psychiatric medication (including antidepressants, antipsychotics and antiepileptic drugs)
* Youths who have limited comprehension due to epilepsy or mental retardation.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in psychological distress | Baseline, 3-month, 6-month, and 1 year
  Distress item from Kessler-6 (K-6), scores range from 0-24, higher scores indicate higher distress level

SECONDARY OUTCOMES:
Change in depressive and anxiety | Baseline, 3-month, 6-month, and 1 year
  Depression and Anxiety subscales in Depression Anxiety Stress Scales (DASS), scores range from 0-42, higher scores indicate higher symptom level
Change in functioning | Baseline, 3-month, 6-month, and 1 year
  Productivity loss (1-item in K6) and Social and Occupational Functioning Assessment Scale (SOFAS), scores range from 0-100, higher scores indicate better functioning

CONTACTS AND LOCATIONS:
Overall Officials: Eric Yu Hai Chen, FHKAM(Psychiatry), Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Psychiatry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hui CL, Suen YN, Lam BY, Wong SM, Wong CS, Lui SS, Chan KT, Wong MT, Chan SK, Lee EH, Chang WC, Wong GH, Chen EY. LevelMind@JC: Development and evaluation of a community early intervention program for young people in Hong Kong. Early Interv Psychiatry. 2022 Aug;16(8):920-925. doi: 10.1111/eip.13261. Epub 2021 Dec 11. PMID 34894378